CLINICAL TRIAL: NCT05404672
Title: Effects Of Breathing Exercises With And Without Aerobic Training On Dysfunctional Breathing And Exercise Intolerance In Patients With Postural Orthostatic Tachycardia Syndrome
Brief Title: Breathing Exercises With And Without Aerobic Training In Patients With Postural Orthostatic Tachycardia Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR&AHS/22/0320
Record Dates: First submitted 2022-05-31; First posted 2022-06-03 (Actual); Last update posted 2023-01-25 (Actual); Status verified 2023-01

CONDITIONS: Postural Orthostatic Tachycardia Syndrome
Keywords: Postural orthostatic tachycardia syndrome; Dysfunctional Breathing; Aerobic Training; Exercise Intolerance; Progressive Breathing Retraining
MeSH Terms: conditions — Postural Orthostatic Tachycardia Syndrome

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aerobic Training (Experimental): Progressive breathing training exercises for a period of 4 weeks, for 15 minutes twice daily. As patients progressed to the seated posture, the controlled pause technique (exercise) will be introduced. 4 times a day followed by a sustained period of breathing control. In addition to this Aerobic Training (cycling, treadmill) will also be practiced for 30 minutes constituting 5 days/ week. Initial training would avoid upright position. Mild-to-moderate-intensity endurance training, progressing from semi-recumbent to upright position plus strength training will be practiced.
  Interventions: Other: Aerobic Training; Other: Conventional Treatment
- Conventional Treatment (Active Comparator): Progressive breathing retraining exercises for a period of 4 weeks, for 15 minutes twice daily. As patients progressed to the seated posture, the controlled pause technique (exercise) will be introduced. 4 times a day followed by a sustained period of breathing control.
  Interventions: Other: Conventional Treatment

INTERVENTIONS:
Other: Aerobic Training — Progressive breathing retraining exercises for a period of 4 weeks, for 15 minutes twice daily. As patients progressed to the seated posture, the controlled pause technique (exercise) will be introduced. 4 times a day followed by a sustained period of breathing control. In addition to this Aerobic Training (cycling, treadmill) will also be practiced for 30 minutes constituting 5 days/ week. Initial training would avoid upright position. Mild-to-moderate-intensity endurance training, progressing from semi-recumbent to upright position plus strength training will be practiced.
  Arms: Aerobic Training
Other: Conventional Treatment — Progressive breathing retraining exercises for a period of 4 weeks, for 15 minutes twice daily. As patients progressed to the seated posture, the controlled pause technique (exercise) will be introduced. 4 times a day followed by a sustained period of breathing control.

SUMMARY:
Postural orthostatic tachycardia syndrome (POTS) is a chronic, multifactorial syndrome with complex symptoms of orthostatic intolerance. Of the major complaints are breathlessness and exercise intolerance. The aim is to explore the potential impact of a physiotherapy intervention involving education and breathing control on dysfunctional breathing and improving exercise intolerance in POTS. The study would be a randomised controlled trial. Duration would be 4 week. Patients will be randomly divided into two groups by lottery method. Data will be collected through questionnaire from enrolled subjects in physical therapy department of Liaqat Hospital, Lahore. Experimental group will be treated by Progressive Breathing Retraining Exercise Program-2 times a day for 15 minutes, initially Controlled Nasal Breathing with progressively increasing the Controlled Pause, 4 times a day for 15 minutes, then both techniques will be performed together. In addition to this Aerobic training will be assigned to both the groups. Aerobic training will include cycling and treadmill- for 30 minutes\day for 5 days\week for 1 month. Total 20 sessions. While the controlled group will receive only aerobic training which will include cycling and treadmill for 30 minutes\day for 5 days\week for 1 month. Total 20 sessions. The dysfunctional breathing and exercise intolerance will be assessed through Nijmegen Questionnaire and Veterans Questionnaire respectively at 0 week, after 2 week and after 4 week. The data will be analyzed by spss version 25.

ELIGIBILITY:
Inclusion Criteria:

* Only Females
* Age: (15-45years)
* +ve tilt table test
* +ve 10 minutes standing test
* Nijmegen score >22,
* increase in HR>30bpm; with no orthostatic fall in blood pressure.symptoms occuring in >3 months

Exclusion Criteria:

* pregnancy
* No cardiac or respiratory pathology
* Surgical history
* Participants in another research protocol
* Any other medical condition that confers greater morbidly than POTs (e.g.,active Cancer)

Ages: 15 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes
Enrollment: 28 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-01-15 (Actual)

PRIMARY OUTCOMES:
Nijmen Questionnaire ….dysfunctional breathing | 4 week.
  This questionnaire is a self-report 16-symptom scale. The frequency of symptoms can be indicated by the following options (score): never (0), rarely (1), sometimes (2), often (3), and very often (4). This questionnaire was developed to screen individuals complaining of shortness of breath with several signs and symptoms of hyperventilation syndrome, such as tense feeling, dizziness, fast and deep breathing, feeling of tightness around the mouth, and anxiety.
  Readings will be at 0 week, after 2 week and after 4 week
Veterans specific activity questionnaire (VSAQ): | 4 week
  The Veterans Specific Activity Questionnaire (VSAQ) is a 13-item self-administered symptom questionnaire that estimates aerobic fitness expressed in metabolic equivalents (METs). Aerobic capacity is measured in METs by the VSAQ.
  Readings will be at 0 week, after 2 week and after 4 week

CONTACTS AND LOCATIONS:
Overall Officials: Hafiza Muriam Ghani, MSPT-CP, Principal Investigator — Riphah International University
Locations (1):
- Liaqat Hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Abed H, Ball PA, Wang LX. Diagnosis and management of postural orthostatic tachycardia syndrome: A brief review. J Geriatr Cardiol. 2012 Mar;9(1):61-7. doi: 10.3724/SP.J.1263.2012.00061. PMID 22783324
- [Background] Reilly CC, Floyd SV, Lee K, Warwick G, James S, Gall N, Rafferty GF. Breathlessness and dysfunctional breathing in patients with postural orthostatic tachycardia syndrome (POTS): The impact of a physiotherapy intervention. Auton Neurosci. 2020 Jan;223:102601. doi: 10.1016/j.autneu.2019.102601. Epub 2019 Nov 12. PMID 31743851
- [Background] Deb A, Morgenshtern K, Culbertson CJ, Wang LB, Hohler AD. A survey-based analysis of symptoms in patients with postural orthostatic tachycardia syndrome. Proc (Bayl Univ Med Cent). 2015 Apr;28(2):157-9. doi: 10.1080/08998280.2015.11929217. PMID 25829642
- [Background] Jarosz B. POSTURAL ORTHOSTATIC TACHYCARDIA SYNDROME (POTS): ITS RELEVANCE, AND IMPORTANCE, IN THE MANAGEMENT OF SPORT RELATED CONCUSSION. Chiropractic Journal of Australia. 2021;48(1):31-4.
- [Background] Raj SR, Guzman JC, Harvey P, Richer L, Schondorf R, Seifer C, Thibodeau-Jarry N, Sheldon RS. Canadian Cardiovascular Society Position Statement on Postural Orthostatic Tachycardia Syndrome (POTS) and Related Disorders of Chronic Orthostatic Intolerance. Can J Cardiol. 2020 Mar;36(3):357-372. doi: 10.1016/j.cjca.2019.12.024. PMID 32145864
- [Derived] Dani M, Fedorowski A. Tackling POTS Needs More Than Just a Sympathetic Approach. Hypertension. 2024 Nov;81(11):2248-2250. doi: 10.1161/HYPERTENSIONAHA.124.23716. Epub 2024 Oct 16. No abstract available. PMID 39413203